CLINICAL TRIAL: NCT01959217
Title: Targeting Prospective Memory to Improve HIV Adherence in Adolescents at Risk for Substance Abuse
Brief Title: Targeting PM to Improve HIV Adherence in Adolescents at Risk for Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Angulique Outlaw, Associate Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA034497 (NIH)
Record Dates: First submitted 2013-08-30; First posted 2013-10-09 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Adherence; Substance Abuse
Keywords: HIV; Substance Abuse; Prospective Memory
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PM Component Text Reminders (Experimental): There will be a a single face-to-face intervention followed by tailored text reminders. The number of PM components (strategic encoding, monitoring, and cue salience) that will comprise the tailored text message reminders will be determined by Phase 1.
  Interventions: Behavioral: PM Component Text Reminders

INTERVENTIONS:
Behavioral: PM Component Text Reminders — The number of PM components (strategic encoding, monitoring, and cue salience) that will comprise the tailored text reminders will be determined by Phase 1.

SUMMARY:
Medication adherence rates among youth living with HIV are inadequate to effectively manage the disease, and novel interventions grounded in basic behavioral sciences are needed. This multi-site phased (3 phases) study plans to translate basic cognitive neuroscience regarding prospective memory (PM) into a more potent adherence intervention for youth living with HIV (YLH).

The phases are:

Phase 1: To improve PM in basic laboratory tasks in YLH with and without substance abuse.

-Hypothesis 1: Manipulations in three theory-based components of PM (strategic encoding, self-monitoring and cue salience) will improve PM within each participant.

Phase 2: To conduct proof of concept studies of a text-delivered PM intervention for taking ART in YLH with suboptimal adherence.

* Hypothesis 2: Using a multiple baseline across subjects design, adherence to antiretroviral therapy (ART) will improve following initiation of the PM adherence intervention and will be maintained for 6 weeks after tapering of the intervention.
* Hypothesis 2a: Similar feasibility, tolerability, and adherence improvement trends will be seen in youth with and without substance problems.

Phase 3: To conduct additional proof of concept studies, based on Phase 2 findings, of a text-delivered PM intervention for taking ART in YLH with suboptimal adherence.

* Hypothesis 3: Using a multiple baseline across subjects design, adherence to ART will improve following initiation of the PM adherence intervention and will be maintained for 6 weeks after tapering of the intervention.
* Hypothesis 3a: Similar feasibility, tolerability, and adherence improvement trends will be seen in youth.

DETAILED DESCRIPTION:
Medication adherence rates among youth living with HIV are inadequate to effectively manage the disease, and novel interventions grounded in basic behavioral sciences are needed. Emerging evidence suggests that prospective memory (PM) could represent an important piece of the puzzle. PM is defined as the neurocognitive capacity to successfully form, maintain, and execute an intention at a particular point in the future in response to a specific cue. This study plans to translate basic cognitive neuroscience regarding PM into a more potent adherence intervention for YLH, a population at high risk for poor cognitive function, substance abuse, and poor adherence. While text message reminders are an increasingly popular adherence support, evidence of efficacy is equivocal particularly for the maintenance of adherence after reminders end. By using basic cognitive neuroscience to enhance the potency of technology-based interventions to improve PM for adherence tasks, we hope to achieve both greater initial gains as well as sustained improvements in adherence for youth with and without substance abuse.

This multi-site phased study plans to translate basic cognitive neuroscience regarding PM into a more potent adherence intervention for youth living with HIV (YLH).

* In Phase 1, we conducted theory-driven laboratory studies to improve three components of PM using a within-subjects design and traditional cognitive neuroscience tasks (strategic encoding, monitoring, and cue salience) in 60 youth from clinics where the principal investigators (PIs) are located (Detroit and San Diego).
* In Phase 2, we translated promising Phase 1 PM interventions to the youth's natural context, targeting adherence in combination with text messaging, and test for signals of efficacy using a multiple baseline design for YLH with suboptimal adherence (N=24; 12 with substance abuse and 12 without from Detroit).
* In Phase 3, we repeated the Phase 2 study (targeted adherence in combination with text message reminders and two-way assessment text messages, and tested for signals of efficacy using a multiple baseline design for YLH with suboptimal adherence; N=20; Detroit and national online recruitment).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Ability to speak and understand English
* Prescribed antiretroviral therapy for at least 24 weeks
* Detectable viral load in the last month
* Second detectable viral load in the previous 6 months
* Prescribed a regimen with at least two active drugs at study entry
* Regular access to a cell phone with text messaging.

Exclusion Criteria:

* Not fluent in English
* History of severe learning disability, mental retardation, major psychiatric disorders (e.g., schizophrenia, bipolar disorder, major depression with psychotic features, etc.).
* History of a neurological conditions that might influence cognitive functioning (e.g., traumatic brain injury with loss of consciousness > 30 min, central nervous system neoplasms, stroke, seizure disorders, etc.).
* Participation in another adherence intervention trial
* On ART due to pregnancy.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2012-12-13 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Change in Medication Adherence | Change from baseline measurement to 3-months, change from 3-months to 6-months, and change from baseline to 6 months
  Viral load measurement will be obtained by a blood sample to measure medication adherence

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar-King, Ph.D., Principal Investigator — University of Florida; Steven P Woods, Ph.D., Principal Investigator — University of Houston; Angulique Y Outlaw, Ph.D., Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - Wayne State University, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weber E, Blackstone K, Woods SP. Cognitive neurorehabilitation of HIV-associated neurocognitive disorders: a qualitative review and call to action. Neuropsychol Rev. 2013 Mar;23(1):81-98. doi: 10.1007/s11065-013-9225-6. Epub 2013 Feb 16. PMID 23417497
- [Result] Faytell MP, Doyle K, Naar-King S, Outlaw A, Nichols S, Twamley E, Woods SP. Calendaring and alarms can improve naturalistic time-based prospective memory for youth infected with HIV. Neuropsychol Rehabil. 2018 Sep;28(6):1038-1051. doi: 10.1080/09602011.2016.1236733. Epub 2016 Sep 30. PMID 27687290
- [Result] Faytell MP, Doyle KL, Naar-King S, Outlaw AY, Nichols SL, Casaletto KB, Woods SP. Visualisation of future task performance improves naturalistic prospective memory for some younger adults living with HIV disease. Neuropsychol Rehabil. 2017 Dec;27(8):1142-1155. doi: 10.1080/09602011.2015.1122636. Epub 2015 Dec 21. PMID 26690580
- [Result] Woods SP, Doyle KL, Morgan EE, Naar-King S, Outlaw AY, Nichols SL, Loft S. Task importance affects event-based prospective memory performance in adults with HIV-associated neurocognitive disorders and HIV-infected young adults with problematic substance use. J Int Neuropsychol Soc. 2014 Jul;20(6):652-62. doi: 10.1017/S1355617714000435. Epub 2014 May 16. PMID 24834469
- [Result] Loft S, Doyle KL, Naar-King S, Outlaw AY, Nichols SL, Weber E, Casaletto KB, Woods SP. Allowing brief delays in responding improves event-based prospective memory for young adults living with HIV disease. J Clin Exp Neuropsychol. 2014;36(7):761-72. doi: 10.1080/13803395.2014.942255. Epub 2014 Aug 13. PMID 25116075